CLINICAL TRIAL: NCT04263922
Title: Huaiqihuang Granules in the Treatment of Primary Glomerulonephritis of Stage CKD3: a Randomized, Double-blind, Double-simulation, Positive Parallel Control Multi-center Clinical Study
Brief Title: Huaiqihuang Granule in the Treatment of Primary Glomerulonephritis of Stage CKD3
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Collaborators: Huazhong University of Science and Technology (Other); LinkDoc Technology (Beijing) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HQH-201911
Record Dates: First submitted 2019-12-03; First posted 2020-02-11 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-06

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Primary Glomerulonephritis; Huaiqihuang Granule; CKD3
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Valsartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Huaiqihuang group (Experimental): Combine the use of Huaiqihuang granules and Valsartan capsule simulant.
  Interventions: Drug: Huaiqihuang granules
- Valsartan Group (Active Comparator): Combine the use of Valsartan capsule and Huaiqihuang granules simulant.
  Interventions: Drug: Valsartan capsule

INTERVENTIONS:
Drug: Huaiqihuang granules — Huaiqihuang granules, 2 bags at a time, 3 times a day. Valsartan capsule simulant, 80mg at a time, once a day. Oral administration.
  Other Names: B12000050755
  Arms: Huaiqihuang group
Drug: Valsartan capsule — Valsartan capsule, 80mg at a time, once a day. Huaiqihuang granules simulant, 2 bags at a time, 3 times a day. Oral administration.
  Other Names: H20030638
  Arms: Valsartan Group

SUMMARY:
This is a multicentre prospective, randomized, double-blind and imitation, positive-drug parallel controlled clinical trail. The objective of this study is to evaluate the efficacy and safety of Huaiqihuang Granule in patients with CKD stage 3 primary glomerulonephritis.

DETAILED DESCRIPTION:
Chronic kidney disease is a common disease that affects health seriously. In some regions of China, the morbidity of this kind of disease is as high as 10.8%. Primary glomerulopathy is one of the pathogenesis of chronic kidney disease, which occupied 50%-60%. However, at present, there is still a lack of effective means for the treatment of primary glomerulonephritis in CKD stage 3. Huaiqihuang Granule is a kind of Chinese herbal medicine compound preparation, Previous researches showed that Huaiqihuang has a comprehensive effect on primary glomerulonephritis. In this study, there were about 40 first-class hospitals participating in. We planned to enroll 466 participants, who will be randomly divided into the Huaiqihuang Granule group (experimental group) and the Valsartan group (control group). All participants will take medication for 48 weeks, and investigators will follow up participates at weeks 0, 8,16, 24, 32, 40, 48.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as primary glomerulonephritis by renal biopsy
2. Male or female, 18≤age≤65
3. Blood pressure can be effectively controlled at or below 140/90mmHg
4. 30mL/（min.1.73m2）≤ eGFR<60mL/（min.1.73m2）
5. 24-hour urine protein ration ≤ 2.0g/24h
6. The participants must be capable of understanding and comply with the protocol and sign a written informed consent document

Exclusion Criteria:

1. Diagnosed as secondary glomerulonephritis
2. Exposure to corticosteroids, immunosuppressors, tripterygium glycosides, ARBs or ACEIs, without a two weeks washout period
3. Blood pressure < 90/60 mmHg
4. Serum potassium > 5.5 mmol/L
5. Serum albumin < 30g/L
6. Unilateral or bilateral renal artery stenosis
7. Pregnant or lactating women, and participants (including males) who were unable or unwilling to take adequate contraception during the study period
8. Having comorbidities that affect the progression of primary glomerulonephritis (including but not limited to Malignant tumors, Systemic autoimmune diseases, Liver cirrhosis, Diabetes, and Gout)
9. Allergic to the Huaiqihuang Granule or valsartan
10. Participating in another clinical trial
11. Investigators do not think it suitable for a participant to join this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Rate of change in Estimated Glomerular Filtration Rate (eGFR) compared to baseline | 48 weeks
  Events based on eGFR measure compared to baseline calculated using the CKD-EPI formula.

SECONDARY OUTCOMES:
Change in serum creatinine levels from baseline | Start of treatment until the end of the treatment for 48 weeks
  Serum creatinine is being assessed once every 8 weeks for a total of 6 times during the whole study
Change in 24-hour urine protein ration from baseline. | Start of treatment until the end of the treatment for 48 weeks
  Urinary protein is being assessed once every 8 weeks for a total of 6 times during the whole study
Changes in urine erythrocyte levels from baseline | Start of treatment until the end of the treatment for 48 weeks
  Urine erythrocyte is being assessed once every 8 weeks for a total of 6 times during the whole study

OTHER OUTCOMES:
Composite endpoint incidence | Start of treatment until the end of the treatment for 48 weeks
  The incidence of endpoint events：① eGFR decreased by 15% from baseline and was reviewed within 2 weeks, if no improvement was found or if the eGFR continued to decrease by 15% below baseline；② Serum creatinine doubles or enters maintenance of renal replacement therapy or death
Incidence of adverse events | Start of treatment until the end of the treatment for 48 weeks
  The proportion of patients with adverse events to the total population.
Incidence of adverse reactions | Start of treatment until the end of the treatment for 48 weeks
  The proportion of patients with adverse reactions to the total population

CONTACTS AND LOCATIONS:
Overall Officials: Hongli Lin, MD, Principal Investigator — The First Affiliated Hospital of Dalian Medical University
Locations (34):
- China (34):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Hebei North University, Zhangjiakou, Hebei
  - The 2nd Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Provincial people's Hospital, Zhengzhou, Henan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The first affiliated Hospital of Baotou Medical College of Inner Mongolia University of Science and Technology, Baotou, Inner Mongolia
  - Affiliated Hospital of Chifeng University, Chifeng, Inner Mongolia
  - Changzhou NO.2 People's Hospital, Changzhou, Jiangsu
  - Jiangsu Province Hospital of Chinese Medicine, Nanjing, Jiangsu
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Anshan Central Hospital, Anshan, Liaoning
  - Anshan Shuangshan Hospital, Anshan, Liaoning
  - Ansteel Group General Hospital, Anshan, Liaoning
  - Benxi Iron and Steel General Hospital of Liaoning Health Industry Group, Benxi, Liaoning
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Dalian Ruikaier Nephropathy Hospital, Dalian, Liaoning
  - Shengjing Hospital of China Medical University( Huaxiang Area), Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Central Hospital affiliated to Shenyang Medical College, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University (Nanhu Area), Shenyang, Liaoning
  - Yingkou Central Hospital, Yingkou, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The Sixth People's Hospital affiliated to Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiaotong University School of medicine, Shanghai, Shanghai Municipality
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Provincial people's Hospital, Taiyuan, Shanxi
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Kunming Yan'an Hospital, Kunming, Yunnan
  - Zhejiang Provincial people's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided